CLINICAL TRIAL: NCT07042932
Title: Online Physical Activity and Health Counseling for Survivors of Childhood Acute Lymphoblastic Leukemia (OPAC-ALL)
Brief Title: Online Physical Activity and Health Counseling for Survivors of Childhood Acute Lymphoblastic Leukemia
Acronym: OPAC-ALL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Hanne Baekgaard Larsen, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: P-2024-15388
Record Dates: First submitted 2025-06-17; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphoblastic Leukemia ALL; Childhood Cancer Survivors; Exercise; Rehabilitation Exercise
Keywords: Exercise; rehabilitation; Acute lymphoblastic leukemia; childhood cancer survivors
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled trial with primary outcome of 26 weeks of exercise. Following primary outcome assessment, the control will receive the intervention components.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (No Intervention): This arm will receive institutional follow-up care during the first 26 weeks. afterward they will receive the intervention
- Exercise (Other): the intervention group will receive 26 weeks of online supervised exercise (1-2 sessions per week) + access to an 8 modele educational material on a webpage + weekly motivational counseling sessions
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — 26 weeks online high intensity functional training, performed 1-2 times per week + access to a LIFESTYLE PHYSICAL ACTIVITY WEBSITE including 8 modules; 1) Welcome, information about the intervention and the aims of the study, 2) Living a physically active lifestyle, 3) Sedentary behavior, 4) General exercise recommendations, 5) How to stay motivated, 6) Strength training, 7) flexibility, balance, and coordination, and 8) Healthy eating + weekly motivational counseling
  Arms: Exercise

SUMMARY:
Advances in the medical treatment of childhood acute lymphoblastic leukemia (ALL) have resulted in 5-year survival rates above 90%- however, the success is not without consequences. Childhood ALL survivors experience markedly impaired physical capacity - reducing their opportunity to engage in everyday activities including leisure activities, sports, and school - affecting their quality of life. Furthermore, Childhood ALL survivors have markedly increased risk of chronic medical conditions including cardiometabolic diseases - that can be prevented through an active lifestyle. Thus, it is imperative to develop novel interventions that can mitigate these treatment-related late-effects. In this RCT, including 82 childhood ALL survivors (10-21 years-old), we will investigate a 26-week online exercise intervention combined with access to a lifestyle physical activity webpage, and health consultations on cardiorespiratory fitness (primary outcome) markers of metabolic syndrome, and physical activity habits.

While other pilot studies have investigated the effects of exercise for childhood ALL survivors, this study is the first RCT internationally to investigate the effects of online exercise combined with education through an app and health counselling for childhood ALL survivor. Using this approach, we are geographically able to reach every survivor in our targeted population, thereby, minimizing logistic challenges like travel distances.

This study has the potential to radically change the way physical rehabilitation is approached in childhood ALL survivors - Potentially changing the workflow of health professionals from referring only survivors with specific deficits to local physiotherapy to referring all survivors to an exercise program tailored to their needs. By improving the children's general physical capacity, we can give the children the required tools to re-enter everyday life activities, including school physical education, leisure activities, and sports earlier after treatment has ended - ultimately minimizing the social complications of treatment. This study will also answer the government´s call to digitalize 30% of rehabilitation by the 2030.

ELIGIBILITY:
Inclusion Criteria:

* aged 10-21 years old,
* at least one year from ended treatment of acute lymphoplastic leukemia
* not adhering to WHO's recommendations for physical activity (i.e., 60 minutes of daily moderate-to-vigorous intensity physical activity including two weekly sessions of strength training for children and 150 minutes of moderate-to-vigorous intensity weekly for adults),
* followed at the pediatric oncology out-patient clinic at Copenhagen University Hospital, Rigshospitalet.

Exclusion Criteria:

* Children with a mental disability,
* other severe physical co-morbidity contradicting physical exercise,
* and/or terminal illness

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
cardiorespiratory fitness (VO2peak (ml/min/kg) | at enrollment and 26 weeks after inclusion
  The primary outcome is the difference in cardiorespiratory fitness (VO2peak (ml/min/kg)) between the intervention group and the waiting list control group after 26- weeks.
  VO2peak is defined as the highest mean over 30 s and expressed in mL/kg/min
  Furthermore, two objective criteria need to be fulfilled before the test is valid. The criteria are heart rate >85% of estimated maximal heart rate and a respiratory exchange ratio (RER)>1.1.

SECONDARY OUTCOMES:
Physical activity and sedentary time | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year- post intervention assessment
  Physical activity and sedentary time are assessed by accelerometers worn for 7 days. The accelerometers (ActiGraph™ model GT3X+, ActiGraph LLC, Pensacola FL, USA) measures accelerations of ±6 G. The sample rate will be set to measure raw signals at 100 Hz, translated into metabolic energy equivalents of light, moderate and vigorous physical activity, and sedentary time. The validity of the Actigraph accelerometer is good, with correlations of 0.65 between accelerometer assessed metabolic energy equivalents and indirect calorimetry Further, we will investigate whether international guidelines for physical activity are met according to established cut-off levels.
cardiorespiratory fitness (VO2peak (ml/min/kg) | at 52 weeks after inclusion and 1-year post intervention
  The primary outcome is the difference in cardiorespiratory fitness (VO2peak (ml/min/kg)) between the intervention group and the waiting list control group after 26- weeks.
  VO2peak is defined as the highest mean over 30 s and expressed in mL/kg/min
  Furthermore, two objective criteria need to be fulfilled before the test is valid. The criteria are heart rate >85% of estimated maximal heart rate and a respiratory exchange ratio (RER)>1.1.
Lower extremity isometric knee extension strength: | at enrolment, 26-weeks after inclusion, 52 weeks after inclusion, 1-year post intervention
  Isometric leg extension is tested using a special-build strength ergometer (Gym 2000®) with a dynamometer (US2A100 kg, Holtinger, Germany) and amplifier. Data is collected through an AD-card (100 HZ) with customized software (LabVIEW ®, National Instruments, Texas, USA). Each participant receives detailed instructions on how to perform each test and is given time to familiarize with each test to secure valid measures.
  The participant is instructed to kick (forward) with maximal force and is obligated to keep maximal intensity for at least five seconds. Three attempts with a two-minute break is carried out, however the participant can try as many attempts as possible if the participant keeps showing improvements. The highest score is noted.
Handgrip strength: | at enrolment, 26 weeks after inclusion, 52 weeks after inclusion 1 year post intervention
  Handgrip strength is measured using a hand-held dynamometer. Participants are placed in a seated position with the elbow flexed at 90°, with three attempts performed for each hand. During testing, the participant will be encouraged to exhibit the best possible force, and the best measure in the strongest hand will be used as test score.
Maximal Leg extension power: | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  Maximal voluntary muscle force will be measured from both legs following a fixed protocol. Leg extensor power will be measured using an extension Power Rig (Nottingham Power Rig, Queen's Medical Centre Nottingham, NG7 2UH, United Kingdom), with subjects positioned with joint angles as if the participant was rising from a chair. Participants are carefully instructed to keep their hands across the chest and to not move the upper body while pushing. Verbal encouragement will be given to ensure maximal performance. The participants extend one leg as forcefully as possible, and the velocity of the flywheel is measured by an opto-switch and used to calculate average leg extensor power in the push. Dominant leg will be tested, a minimum of 5 attempts is carried out for each leg, however the participant continues until two attempts are lower than the maximum (50). The result is expressed in watt (W).
Body arthrometric: | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  Height (m) will be assessed without shoes to the nearest 0.1 cm. Weight (kg) will be measured (no shoes, with underwear or light clothing) to the nearest 0.1 kg and subsequently body mass index (BMI) will be calculated (kg/m2).
Waist circumference | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  Waist circumference will be measured around the abdomen at the level of the umbilicus (cm)
Quality of Life questionnaire | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  The Pediatric Quality of Life Inventory (PedsQL Core) [44] measures the quality of life in children using 23 items on a five-point response scale from never to almost always. The answers are divided into four domains: health and physical activity, emotions, dealing with others, and school activity.
Fatigue/quality of life - PedsQL Multidimensional Fatigue Scale | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  Composed of 18 items, the PedsQL Multidimensional Fatigue Scale [44] possesses three subscales: general fatigue, sleep and rest fatigue, and cognitive fatigue.
Prevalence of Metabolic syndrome: | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  Metabolic syndrome is based on waist and hip circumference, BMI, triglycerides, total cholesterol, high-density lipoprotein (HDL) cholesterol and low-density lipoprotein (LDL) cholesterol, blood pressure, fasting blood sugar and insulin; Within these parameters the International Diabetes Foundation (IDF)
  Blood samples will be obtained following an overnight fast, measuring serum insulin, glucose, total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, total cholesterol, and triglyceride levels. We will collect 15-20 ml per blood sample, (maximum of 2 ml/kg/day including the volume taken for routine clinical analysis). Blood samples will be drawn from an antecubital vein.
  In accordance with the WHO recommendations, no more than 2 ml/kg/day will be drawn and a maximum of 20mL (5). Local anesthetics cream will be used to minimize pain.
  in mmol/L
hip circumference | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  Hip circumference (in CM) at a level parallel to the floor, at the largest circumference of the buttocks following standards described by the World Health Organization. Metabolic syn-drome is based on age-based criterias defined by the International Diabetes Foundation
Body Mass Index | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  Weight and Height is combined to report BMI in kg/m^2
Body composition: Fat-Free Mass | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  Fat-Free Mass (kg and %) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body
Body composition- Bone Mineral Density | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  Bone Mineral Density (g/cm2) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body
Body composition: Bone Mineral Content | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  Bone Mineral Content (kg) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Corporation Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body.
Body composition: Body Fat | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  Body Fat (kg and %) will be analyzed by whole-body DXA scan (DPX-IQ) (Lunar, Lunar Cor-poration Madison, WI, USA). Transverse scans at 1 cm intervals are made from head to toe measuring the absorption of x-ray beams at two different energy levels as these are sent through the body

OTHER OUTCOMES:
Qualitative evaluation of the interventions | at 26 weeks after inclusion
  Experienced project members will conduct semi-structured, in-depth interviews of children and parents (interviewed separately) to understand factors that can influence an individual's likelihood of engaging in physical activity and their perceived experience with participating in the project. Moreover, the feasibility of the intervention components (i.e., online physical activity program, health counseling, lifestyle physical activity website, and education of local trainers) will be explored qualitatively. Furthermore, the health counseling sessions will be recorded.
  Analysis: All data will be transcribed and analyzed according to principles of pragmatic thematic analysis (semi-structured in-depth interviews) or content analysis (recording of health counseling sessions).
General Physical Acivity: Self-Report | at enrollment, 26 weeks after inclusion, 52 weeks after inclusion, 1 year post intervention
  An validated questionnaire used in the UNGkan and HEIA project will be used to assess self-reported physical activity, physical function, sedentary time, screen time, diet habits, active transportation behavior, physical education participation, perceived barriers/facilitators to physical activity, health-related behaviors. The questionnaire contains 35 items

CONTACTS AND LOCATIONS:
Overall Officials: Martin K Fridh, Ph.D, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: Yes
following the final analyses of the study, the IPD will be available upon request
Supporting Information: Study Protocol, SAP